CLINICAL TRIAL: NCT05051475
Title: Endoscopic Radiofrequency Ablation Versus Hybrid Argon Plasma Coagulation in the Treatment of Barrett's Esophagus - the Patients' Perspective: a Randomized Controlled Trial Assessing Procedural Acceptability and Safety (RATE Study)
Brief Title: Endoscopic Radiofrequency Ablation Versus Hybrid Argon Plasma Coagulation in the Treatment of Barrett's Esophagus
Acronym: RATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-21 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-05

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma; Reflux Disease
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- radiofrequency ablation (Active Comparator): Circumferential ablation with radiofrequency ablation will be performed for each segment of the BE starting from the proximal end with one ablation at 12J/cm2, followed by cleaning of mucosal slough with esophageal cap, patient extubation, cleaning of ablation device with wet gauze, and finally a second ablation at 12 J/cm2 (1 × 12J/cm2-clean-1 × 12 J/cm2). Focal ablations will be performed with three consecutive ablations at 12 J/cm2 without cleaning (simplified protocol).
  Interventions: Procedure: Endoscopic radiofrequency ablation
- hybrid argon plasma coagulation (Active Comparator): Patients in the Hybrid argon plasma coagulation group will be treated with a single ablation per session with a power limitation of 60 W (pulsed mode (VIO® 300 D & APC 2, PULSED APC®, Effect 2). No scraping with the endoscope cap and second ablation will be performed.
  Interventions: Procedure: Endoscopic hybrid argon plasma coagulation

INTERVENTIONS:
Procedure: Endoscopic radiofrequency ablation — Endoscopic ablation technique for Barrett's epithelium
  Arms: radiofrequency ablation
Procedure: Endoscopic hybrid argon plasma coagulation — Endoscopic ablation technique for Barrett's epithelium
  Arms: hybrid argon plasma coagulation

SUMMARY:
This study compares patients' acceptability and safety of two established endoscopic methods for treating dysplastic Barrett's esophagus: radiofrequency ablation versus hybrid argon plasma coagulation.

DETAILED DESCRIPTION:
Both endoscopic radiofrequency ablation (RFA) and argon plasma coagulation (APC) are established treatment modalities for dysplastic Barrett's esophagus. Recently, a modification of the APC method has emerged, which involves a submucosal injection of saline preceding the thermal ablation (hybrid-APC; h-APC). This allows to increase the procedure's safety and presumably reduces the patients' post-procedural discomfort. Although both RFA and h-APC are characterized by high effectiveness in eradicating Barrett's segments, limited data compares the patient-related aspects of the procedures. To fill this knowledge gap, we set out a single-center randomized-controlled trial to compare procedural acceptability, safety, and impact on the quality of life, of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 18 years
* Histologically and endoscopically proven Barrett's esophagus requiring ablation therapy according to the current guidelines
* General health status sufficient to perform an endoscopic procedure (ASA I-III)

Exclusion Criteria:

* Primary or secondary coagulopathy, with INR>1.5 and/or platelet count of <75,000.
* Anticoagulation therapy (e.g. warfarin) for high-risk condition and unable to withhold the medication temporarily
* Recent myocardial infraction or other significant cardiovascular event within 6 months prior to recruitment
* Patients under long-term care and/or within nursing facilities (e.g. psychosocial disorders, mental retardation)
* Any history of esophageal resection surgery
* Esophageal varices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Level of post-procedural pain | Measured at any time point before given anesthesia for the procedure and immidietly after the procedure.
  Change in chest pain evaluated by the numeric analog scale (NAS) from score 0 (no pain) to 10 (worst possible pain) before the procedure and immidietly after (30-60 minutes) the procedure.
Level of post-procedural pain at day 7 after treatment | Measured at day 7 after the procedure
  Post-procedural chest pain evaluated by the numeric analog scale (NAS) from score 0 (no pain) to 10 (worst possible pain)
Level of late post-procedural pain (at day 30 after treatment) | Measured at day 30 after the procedure
  Post-procedural chest pain evaluated by the numeric analog scale (NAS) from score 0 (no pain) to 10 (worst possible pain)

SECONDARY OUTCOMES:
Level of post-procedural dysphagia | Measured before the procedure, immidietly after (30-60mins), and at day 7, and day 30 after the procedure.
  Evaluated by the Mellow-Pinkas scoring from 0 (able to eat normal diet / no dysphagia) to 4 (unable to swallow anything / total dysphagia)
Level of post-procedural quality of life | Measured before the procedure, immidietly after (30-60mins), and at day 7, and day 30 after the procedure.
  Evaluated by the QLQ-OES18 questionnaire specific for esophageal symptoms, and consists of a symptom scale only. The QLQ-OES18 includes 18 questions: 6 single item subscales relating to saliva swallowing, choking, dry mouth, taste, coughing, and talking. It also includes 12 items grouped into 4 subscales: dysphagia (3 items), eating (4 items), reflux (2 items), and pain (3 items).
The rate of complications | Measured during the prcoedure, immidietly after the procedure and at day 7 and day 30 after the procedure during follow-up
  Intra-procedural complications, such as bleeding, perforation, post-procedural complications, e.g. chest-pain, esophageal stricture will be monitored during the hospital stay and follow-up at day 7 and day 30 after the procedure (phone call).

CONTACTS AND LOCATIONS:
Overall Officials: Wladyslaw Januszewicz, MD, Principal Investigator — Centre for Postgraduate Medical Education
Locations (1):
- Medical Centre for Postgraduate Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No